CLINICAL TRIAL: NCT03463005
Title: Male Infertility and Complementary Treatment
Brief Title: The Effect of Royal Vaginal Gel Compared to IUI Technique on Fertility Rate of Women With Low-fertility Husbands
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gonabad University of Medical Sciences (Other)
Collaborators: Mashhad University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Narjes Bahri, Dr Narjes Bahri, Gonabad University of Medical Sciences
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 921175
Record Dates: First submitted 2018-02-18; First posted 2018-03-13 (Actual); Last update posted 2018-03-13 (Actual); Status verified 2018-03

CONDITIONS: Asthenozoospermia
MeSH Terms: conditions — Asthenozoospermia | interventions — royal jelly

STUDY DESIGN:
Intervention Model Description: The study subjects were voluntarily assigned to royal gel and IUI groups. In royal gel group, 5 grams of royal gel was used after menstruation and every other night before and after intercourse. IUI group received 75 units of FSH from the second day of the cycle.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Royal jelly (Experimental): The study subjects included healthy women who had husbands with male-factor infertility problems.
  Interventions: Other: Royal jelly
- IUI group (Active Comparator): The study subjects included in IUI group were healthy women who had husbands with male-factor infertility problems.
  Interventions: Procedure: IUI

INTERVENTIONS:
Other: Royal jelly — The study subjects in the Royal jelly group used 10 ml of the vaginal Royal jell few minutes before and few minutes after intercourse one day after the end of menstruation for two weeks.
  Other Names: Complementary group
  Arms: Royal jelly
Procedure: IUI — Subjects in IUI group received 75 units of FSH from the second day of the cycle.
  Arms: IUI group

SUMMARY:
The present Pocock clinical trial study was conducted In the city of Mashhad in Iran between 2015 and 2016. The study inclusion criteria were men with low fertility of sperm motility<25% and total motility <50% (asthenozoospermia), no history of endocrine diseases, no diabetes men, no hormonal problems in their wives, and a healthy salpingography in their wives. The study subjects were voluntarily assigned to royal gel and IUI groups. In royal gel group, 5 grams of royal gel was used after menstruation and every other night before and after intercourse. IUI group received 75 units of FSH from the second day of the cycle. Then vaginal ultrasound was performed from the sixth day of menstrual cycle to determine the right size of follicle. 10000 units of HCG was administered when follicle diameter reached 16mm, and the study subject was prepared for IUI 32-36 hours later. Each subject alternately swapped groups following fertility failure.

DETAILED DESCRIPTION:
After selection of subjects and obtaining their informed consents, the quality of royal gel was examined.

The quality of royal gel is determined by the amount of polyphenol it contains. Polyphenol in royal gel was assessed in the following stages: first, the sample was diluted with ethanol 50% to 1:10 ratio, and then, 100µl of this preparation was poured into a test tube, and 750µl of 1:10 diluted solution of FCR (Folin Ciocalteau Reagent) was added and left at room temperature for five minutes. Then, 750µl of sodium carbonate 6% solution was added to each tube, and after keeping these tubes in the dark for one hour, absorption was measured at 780nm wavelength. Negative control consisted of all reaction compounds, except the sample, for which, ethanol 50% was used instead. The sample concentration was determined using the gallic acid standard. By definition, the desirable quality of polyphenol in natural royal gel ranges from 0.15mg (minimum) to 0.75mg (maximum) in every 100 grams, and this was determined 0.5 mg for the sample used in the present study, indicating a good quality (15).

ELIGIBILITY:
Inclusion Criteria:

* Male-factor infertility (defined as total sperm motility<40% and sperm motility<20%)
* Normal hormonal profile in women
* Normal hysterosalpingography report
* Regular sexual relationships

Exclusion Criteria:

* Ovulation dysfunction
* History of sexually transmitted diseases in women and men
* Hormonal disorders in men and women

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2017-09-20 (Actual); Study Completion 2017-12-10 (Actual)

PRIMARY OUTCOMES:
Occurrence of pregnancy | Three months after intervention
  Occurrence of pregnancy be detected by B-HCG test

SECONDARY OUTCOMES:
confirmation of pregnancy | Three months after intervention
  Abdominal sonography to approve pregnancy and visit embryo sac.

CONTACTS AND LOCATIONS:
Overall Officials: Tahereh Fathi Najafi, Instructor, Study Director — Midwifery department, Islamic Azad Medical University, Mashhad branc, Mashhad, Iran

IPD SHARING:
Plan to Share IPD: No